CLINICAL TRIAL: NCT04923906
Title: Efficacy and Safety of Aumolertinib with or Without Chemotherapy As First-line Treatment in Locally Advanced or Metastatic Non-Small Cell Lung Cancer with Sensitizing Epidermal Growth Factor Receptor Mutations: a Randomized, Controlled, Open-label, Phase 3 and Multicenter Clinical Study
Brief Title: Aumolertinib with or Without Chemotherapy As 1st Line Treatment in Locally Advanced or Metastatic Non-Small Cell Lung Cancer with Sensitizing EGFR Mutations
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10296-306
Record Dates: First submitted 2021-06-10; First posted 2021-06-11 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Concurrent Chemotherapy, Aumolertinib, EGFR-TKI, EGFRm+, Ex19Del, L858R, HS-10296, Stage IIIB-IV, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aumolertinib and platinum-based chemotherapy (Experimental)
  Interventions: Drug: Aumolertinib
- Aumolertinib (Active Comparator)
  Interventions: Drug: Placebo Aumolertinib

INTERVENTIONS:
Drug: Aumolertinib — Aumolertinib 110 mg QD in combination with pemetrexed (500 mg/m2) plus cisplatin (75 mg/m2) or carboplatin (AUC5) on Day 1 of every 21-day cycles up to 4~6 cycles, followed by Aumolertinib 100mg QD with pemetrexed maintenance (500 mg/m2) on Day 1 of every 21-day cycles.
  Dose may be reduced to allow for the management of investigational drug related toxicity.
  Other Names: HS-10296
  Arms: Aumolertinib and platinum-based chemotherapy
Drug: Placebo Aumolertinib — Placebo Aumolertinib 110 mg QD Dose may be reduced to allow for the management of investigational drug related toxicity.
  Arms: Aumolertinib

SUMMARY:
To assess the efficacy and safety of Aumolertinib plus chemotherapy versus Aumolertinib alone as first-line treatment in locally advanced or metastatic non-small cell lung cancer (NSCLC) with sensitizing epidermal growth factor receptor mutations (EGFRm+).

DETAILED DESCRIPTION:
HS-10296-306 is a randomized, open-label, multicenter, phase III study to assess the efficacy and safety of Aumolertinib plus chemotherapy versus Aumolertinib alone as first-line treatment in locally advanced or metastatic non-small cell lung cancer (NSCLC) with sensitizing epidermal growth factor receptor mutations (EGFRm+). Eligible patients are randomized to receive either Aumolertinib (110 mg orally, once daily) in combination with platinum-based chemotherapy (every 3 weeks for 4~6 cycles) or Aumolertinib (110 mg orally, once daily) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of informed consent before any study-specific procedures, sampling and analyses.

  2. Male or female, age at least 18 years. 3. Histologically confirmed locally advanced or metastatic NSCLC (included patients with stage IIIB, IIIC or IV disease who had relapsed after prior surgery or were newly diagnosed). Patients must be treatment-naïve for locally advanced or metastatic NSCLC. Prior adjuvant and neo-adjuvant therapies are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.

  4. The tumor harbors 1 of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations assessed by central testing using tumor tissue sample or blood sample.

  5. At least 1 lesion that has not previously been irradiated, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm).

  6. An Eastern Cooperative Oncology Group (ECOG) performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.

  7. Female patients should be using adequate contraceptive measures and should not be breastfeeding at the screening period, during the study, and six months after the last dosing of study. Patient must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at screening:
  1. Postmenopausal defined as age more than 50 years and amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments.
  2. Women under 50 years old would be considered postmenopausal if they have been amenorrhea for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
  3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.

     8. Male patients should be willing to use barrier contraception (i.e., condoms).

     Exclusion Criteria:
* 1. Treatment with any of the following:

  1. Prior treatment with an EGFR TKI.
  2. Major surgery (excluding placement of vascular access) within 4 weeks of randomization.
  3. Radiotherapy to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of randomization.
  4. Spinal cord compression or brain metastases unless asymptomatic, stable for at least 4 weeks, and not requiring steroids for at least 2 weeks prior to start of study treatment.
  5. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.

     2. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 at the time of starting study treatment.

     3. History of other malignancies, excluding full treated non-melanoma skin cancer, in-situ cancer, or other solid tumors that hadn't recurrent for > 5 years following the end of treatment.

     4. Inadequate bone marrow reserve or organ function. 5. Any of the following cardiac criteria:

  <!-- -->

  1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) < 50%. 6. Any evidence of severe or uncontrolled systemic diseases (including uncontrolled hypertension and active bleeding diatheses) or active infection. Screening for chronic conditions is not required.

     7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Aumolertinib.

     8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.

     9. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.

     10. History of hypersensitivity to any active or inactive ingredient of study drugs (pemetrexed, cisplatin, carboplatin, Aumolertinib) or to drugs with a similar chemical structure or class to Aumolertinib.

     11. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

     12. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.

     13. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) assessed by IRC (Independent Review Committee) | From the time of randomization to disease progression or death, approximately 3 years.
  IRC-PFS is defined as the time from randomization until the date of objective disease progression based on IRC assessment or death (by any cause in the absence of progression). The patients will receive long-term follow-up including chest and abdominal CT every 6 weeks until Week 18, then every 12 weeks and onwards.

SECONDARY OUTCOMES:
ORR (Objective Response Rate) assessed by IRC (Independent Review Committee) | From the time of randomization to the date of first occurrence of complete response (CR) or partial response (PR), approximately 3 years.
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression.
DoR (Duration of response) | From the time of randomization to disease progression or death, approximately 3 years.
  DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
DCR (Disease Control Rate) | From the time of randomization to disease progression or death, approximately 3 years.
  The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD.
DepOR (Depth of Response) | From the time of randomization to disease progression or death, approximately 3 years.
  DepOR is defined as the sum of the lengths of the longest diameters of the RECIST 1.1 target lesions.
PFS (Progression Free Survival) Rate at 12, 18, 24, and 36 months | The PFS Rate at 12, 18, 24, and 36 months is assessed up to 36 months.
  PFS Rate at 12, 18, 24, and 36 months is defined as proportion of progression free survival at 12, 18, 24, and 36 months from the date of randomization.
OS (Overall survival) | From the time of randomization to death due to any cause, approximately 6 years.
  Overall survival (OS) is deﬁned as the time from randomization to death due to any cause. The survival will be followed up with telephone every 12 weeks after discontinuation of the randomized treatment.
OS (Overall survival) rate at 3, 5 years | The OS rate at 3, 5 years is assessed up to 5 years.
  OS rate at 3, 5 years is defined as the proportion of patients alive at 3, 5 years from the date of randomization.
Incidence and severity of AEs (Adverse Events) | From the screening period to 28 days after treatment completion, approximately 4 years.
  AEs are graded according to CTCAE v5.0 and recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Chest Hospital, China

IPD SHARING:
Plan to Share IPD: No